CLINICAL TRIAL: NCT02222649
Title: EVALUATION OF THE HIGH DOSE VITAMIN D3 SUPPLEMENTATION EFFECT AND INFLUENCE OF POLYMORPHISM VDR GENE ON OXIDATIVE STRESS AND INFLAMMATORY PROCESS IN ELDERLY
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of Paraíba (Other)
Responsible Party: Principal Investigator, Isa G M Cavalcante, DDS, Master student, Federal University of Paraíba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IGabriela; 0374/12 (Other: Federal University of Paraíba Research Ethics Committee of the Center for Health Sciences)
Record Dates: First submitted 2014-08-15; First posted 2014-08-21 (Estimated); Last update posted 2015-03-06 (Estimated); Status verified 2014-08

CONDITIONS: Disorder of Aging
Keywords: Elderly; vitamin D insufficiency; High dose vitamin D3 supplementation; Polymorphism of the VDR gene
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3 (Experimental): Group supplemented with high single dose of 200,000 IU of vitamin D3 (cholecalciferol)
  Interventions: Dietary Supplement: Vitamin D3
- placebo group (Placebo Comparator): Placebo capsules with starch
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — High dose of 200,000 IU of cholecalciferol orally in a single dose
  Other Names: cholecalciferol; High dose
  Arms: Vitamin D3
Dietary Supplement: Placebo — Capsules of starch, no therapeutic action
  Arms: placebo group

SUMMARY:
A vitamin D3 high dose would act as an antioxidant and anti-inflammatory improving markers of oxidative stress and inflammation in the elderly. Seniors exhibiting polymorphism in the VDR gene would become non-responsive to supplementation.

DETAILED DESCRIPTION:
The high prevalence of hypovitaminosis D in the elderly can be identified as a risk factor for developing cardiovascular disease and consequent increase in oxidative stress and chronic inflammation. Polymorphisms in the gene that encodes the vitamin D receptor (VDR) can influence the cellular responses supplementation of vitamin D. The study objective is to evaluate the influence of supplementation of 200,000 in a single high dose of vitamin D3 in the inflammatory status and oxidative stress elderly and the influence of polymorphism of the VDR gene in this response. One randomized, placebo-controlled clinical trial, designed with non-institutionalized elderly in northeastern Brazil will be held. All volunteers will sign the Instrument of Consent and will undergo clinical, nutritional, anthropometric and biochemical evaluation. The purpose is to produce new knowledge helping to unravel the beneficial effects of vitamin D3.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years; diagnosis of failure / vitamin D, preserved cognitive status, disability accepting participate and are not included in any of the exclusion criteria

Exclusion Criteria:

* excluded from the study in the elderly using vitamin D supplements; anticonvulsant drugs or for the treatment of HIV / AIDS; diagnosis of type I diabetes mellitus, nephrotic syndrome, acute or chronic renal failure, liver disease, hypothyroidism, hyperthyroidism, history of cerebrovascular accident (CVA) or acute myocardial infarction (AMI) Vascular past 6 months and chronic consumptive diseases, alcoholic or smoker chronic.

Ages: 60 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-05 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
number of elderly women with sufficient vitamin D levels | four weeks after the intervention

SECONDARY OUTCOMES:
number of elderly who have reduced serum levels of High-Sensitivity C-Reactive Protein | four weeks after the intervention
number of elderly who have reduced serum levels of Alpha 1 Acid Glycoprotein | four weeks after the intervention
number of elderly who have reduced plasma levels of malondialdehyde (MDA) | four weeks after the intervention
number of elderly that increased plasma antioxidant full capacity | four weeks after the intervention

OTHER OUTCOMES:
Number of Participants with Polymorphism of the VDR gene | Participants will be followed for the duration of recruitment , an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Isa Gabriela M Cavalcante, DDS, Principal Investigator — Federal University of Paraíba; Maria da Conceição R Gonçalves, PDH, Study Director — Federal University of Paraíba; Alexandre S Silva, PHD, Study Director — Federal University of Paraíba
Locations (1):
- Program for Attention to Elderly, belonging to the Municipality of João Pessoa, João Pessoa, Paraíba, Brazil